CLINICAL TRIAL: NCT03870217
Title: Comparing Site-selection Strategies for Improving Speech Recognition Outcomes
Brief Title: Comparing Site-selection Strategies
Status: Withdrawn | Type: Observational
Why Stopped: PI passed away. Ending grant and closing lab.
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Heather Wright, Professor, East Carolina University
Other Study IDs: Zhou_R01_study4
Record Dates: First submitted 2019-03-05; First posted 2019-03-12 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness | interventions — Bud13 protein, S cerevisiae

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cochlear implant users with Nucleus and AB devices: Speech recognition will be evaluated after poor electrodes are turned off.
  Interventions: Behavioral: Site selection

INTERVENTIONS:
Behavioral: Site selection — Turning off electrodes on the electrode array based on imaging and psychophysical measures

SUMMARY:
Several studies in the past have tried to deactivate electrodes that are less optimal to improve speech recognition outcomes. The study aims to compare the measures based on which the deactivation was performed. The investigators aim to first examine if the measures are strongly correlated each other, and then compare the deactivation effects across measures. These measures are mainly behavioral including electrode discrimination, amplitude modulation detection thresholds, low-rate and focused detection thresholds and electrode-modiolus distance. The endpoint of the study is speech recognition performance post deactivation.

ELIGIBILITY:
Inclusion Criteria:

* Native speakers of English
* Cochlear Nucleus cochlear implant users or Advanced Bionics users
* Postlingually deafened
* Has had device experience for at least one year
* Can be child or adult at the time of enrollment

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with cochlear implants
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Speech recognition with deactivation | 12 months post award notice and will take up to 3.5 years to complete
  Electrodes will be evaluated based on (1) pitch discrimination (2) focused thresholds (3) amplitude modulation detection thresholds and (4) distances from the modious. Electrodes will be deactivated based on each of these measures and speech recognition will be evaluated to assess the effect of deactivation. The benefit of deactivation (speech recognition after deactivation minus before deactivation) will be derived for each measure. The measure that produces the greatest benefit will be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Zhou, PHD, Principal Investigator — East Carolina University
Locations (1):
- Department of Communication Sciences and Disorders, ECU, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Debruyne JA, Francart T, Janssen AM, Douma K, Brokx JP. Fitting prelingually deafened adult cochlear implant users based on electrode discrimination performance. Int J Audiol. 2017 Mar;56(3):174-185. doi: 10.1080/14992027.2016.1243262. Epub 2016 Oct 19. PMID 27758152
- [Background] Garadat SN, Zwolan TA, Pfingst BE. Using temporal modulation sensitivity to select stimulation sites for processor MAPs in cochlear implant listeners. Audiol Neurootol. 2013;18(4):247-60. doi: 10.1159/000351302. Epub 2013 Jul 20. PMID 23881208
- [Background] Nadol JB Jr. Patterns of neural degeneration in the human cochlea and auditory nerve: implications for cochlear implantation. Otolaryngol Head Neck Surg. 1997 Sep;117(3 Pt 1):220-8. doi: 10.1016/s0194-5998(97)70178-5. PMID 9334769
- [Background] Nadol JB Jr, Young YS, Glynn RJ. Survival of spiral ganglion cells in profound sensorineural hearing loss: implications for cochlear implantation. Ann Otol Rhinol Laryngol. 1989 Jun;98(6):411-6. doi: 10.1177/000348948909800602. PMID 2729822
- [Background] Noble JH, Labadie RF, Gifford RH, Dawant BM. Image-guidance enables new methods for customizing cochlear implant stimulation strategies. IEEE Trans Neural Syst Rehabil Eng. 2013 Sep;21(5):820-9. doi: 10.1109/TNSRE.2013.2253333. Epub 2013 Mar 19. PMID 23529109
- [Background] Seyyedi M, Viana LM, Nadol JB Jr. Within-subject comparison of word recognition and spiral ganglion cell count in bilateral cochlear implant recipients. Otol Neurotol. 2014 Sep;35(8):1446-50. doi: 10.1097/MAO.0000000000000443. PMID 25120196
- [Background] Zhou N. Monopolar Detection Thresholds Predict Spatial Selectivity of Neural Excitation in Cochlear Implants: Implications for Speech Recognition. PLoS One. 2016 Oct 31;11(10):e0165476. doi: 10.1371/journal.pone.0165476. eCollection 2016. PMID 27798658
- [Background] Zhou N. Deactivating stimulation sites based on low-rate thresholds improves spectral ripple and speech reception thresholds in cochlear implant users. J Acoust Soc Am. 2017 Mar;141(3):EL243. doi: 10.1121/1.4977235. PMID 28372106
- [Background] Zhou N, Pfingst BE. Psychophysically based site selection coupled with dichotic stimulation improves speech recognition in noise with bilateral cochlear implants. J Acoust Soc Am. 2012 Aug;132(2):994-1008. doi: 10.1121/1.4730907. PMID 22894220
- [Background] Zwolan TA, Collins LM, Wakefield GH. Electrode discrimination and speech recognition in postlingually deafened adult cochlear implant subjects. J Acoust Soc Am. 1997 Dec;102(6):3673-85. doi: 10.1121/1.420401. PMID 9407659
- [Background] Bierer JA, Litvak L. Reducing Channel Interaction Through Cochlear Implant Programming May Improve Speech Perception: Current Focusing and Channel Deactivation. Trends Hear. 2016 Jun 17;20:2331216516653389. doi: 10.1177/2331216516653389. PMID 27317668
- [Background] Srinivasan AG, Padilla M, Shannon RV, Landsberger DM. Improving speech perception in noise with current focusing in cochlear implant users. Hear Res. 2013 May;299:29-36. doi: 10.1016/j.heares.2013.02.004. Epub 2013 Mar 1. PMID 23467170